CLINICAL TRIAL: NCT03863548
Title: French Observational Study of Complications Associated With Anticoagulants and Antiplatelet Treatment in Retina/Vitreous Surgery (CLOT Study)
Brief Title: French Observational Study of Complications Associated With Anticoagulants and Antiplatelet Treatment in Retina/Vitreous Surgery
Acronym: CLOT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: LOUISON CFSR 2017
Record Dates: First submitted 2019-03-04; First posted 2019-03-05 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Patients Undergoing Retina/Vitreous Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Continuation of antithrombotic drugs: operation carried out without stopping anticoagulants
  Interventions: Other: complication
- Stop anti thrombotic drugs: operation performed with stopping the anticoagulants
  Interventions: Other: complication

INTERVENTIONS:
Other: complication — collection of post-operative bleeding complications

SUMMARY:
Anticoagulants and antiplatelet treatments are frequently prescribed treatments to prevent or treat thromboembolic complications and reduce morbidity and mortality related to cardiovascular risk factors. In retina/vitreous surgery, there are rare but potentially serious risks of hemmorrhagic complication resulting in irreversible loss of visual acuity. There is no clear consensus on how to proceed during the perioperative period with regard to the continuation or discontinuation of anticoagulant and antiplatelet treatments in these types of surgery. the purpose of the study is to identify complications at 1 month depending on the type of surgery with or without discontinuation of antithrombotic treatments. Practitioners are not asked to change their modus operandi. The hypothesis is that there is no excess risk of peri- or post-operative hemorrhage in retino-vitreous surgery in patients treated with antithrombotic compared to untreated patients and that therefore discontinuation of these treatments before surgery is not necessary.

ELIGIBILITY:
Inclusion Criteria:

* person who has expressed willingness to participate
* person over 18 years of age
* person with a retinal-vitreous condition requiring scheduled surgery (epi-retinal membrane surgery, vitreous traction surgery, macular hole surgery).

Exclusion Criteria:

* person subject to legal protection (curatorship, guardianship)
* person deemed mentally incompetent
* pregnant, parturient or breastfeeding woman
* adult unwilling or unable to consent
* patient who has already participated in the study
* person with a physical or mental disability that does not allow participation.
* a person who has participated in any study of an experimental medical product within the previous 3 months
* person who experiences any of the following during the ophthalmological examination:

  * severe or proliferating diabetic retinopathy
  * intra-vitreal hemorrhage
  * tractional retinal detachment
  * subretinal or retrohyaloidal hematoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery
Sampling Method: Non-Probability Sample
Enrollment: 748 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
Occurrence of intra-operative and postoperative hemorrhagic complications in retina/vitreous surgery | Through study completion, an average of 8 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Louison S, Gabrielle PH, Soudry A, Meillon C, Blanc J, Beal G, Arsene S, Le Mer Y, Berrod JP, Kodjikian L, Creuzot-Garcher C; CFCR Research net. Perioperative risk of bleeding with antithrombotic agents in macular surgery: a national, prospective, multicentre study. Acta Ophthalmol. 2020 Dec;98(8):e991-e997. doi: 10.1111/aos.14434. Epub 2020 Apr 12. PMID 32279459